CLINICAL TRIAL: NCT01831297
Title: Haemodynamic Feasibility Study of Sensors Within a Tilting Table Examination
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 10-082
Record Dates: First submitted 2013-01-29; First posted 2013-04-15 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- syncope
  Interventions: Device: measurement of blood pressure

INTERVENTIONS:
Device: measurement of blood pressure — measurement of pulse wave velocity

SUMMARY:
This study´s aim is to explore physiological associations concerning pulse wave velocity, heart rate and blood pressure in order to make taking the blood pressure more comfortable.

ELIGIBILITY:
Inclusion Criteria:

* patients with syncope and planned tilting table investigation
* male and female patients aged at least 18 years
* persons being able to understand and to follow the study stuff´s instructions

Exclusion Criteria:

* pregnancy or breast feeding
* patients not being able to consent
* cardiac pacemaker / defibrillator
* illness of skin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with syncope
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
data about possible correlation | 45 minutes
  Correlation between pulse wave velocity, pulse rate and blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Hospital Aachen, Aachen, North Rhine Westfalia, Germany